CLINICAL TRIAL: NCT02091609
Title: Evaluation of Plaque Removal Using Different Plaque Control Therapies Around Single Crown Dental Implants and Splinted Implant Crowns in Patients Under 3 Months Maintenance;a Randomized Clinical Trial
Brief Title: a Randomized Clinical Trial Evaluating Plaque Removal Around Dental Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H2013:458
Record Dates: First submitted 2014-03-12; First posted 2014-03-19 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2015-05

CONDITIONS: Peri Implantitis
Keywords: plaque removal around dental implants
MeSH Terms: conditions — Peri-Implantitis | interventions — Dental Devices, Home Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group : implants and oral hygiene (Experimental): dental floss
  Interventions: Other: dental floss
- implants and oral hygiene (Experimental): dental interproximal brush
  Interventions: Other: dental interproximal brush

INTERVENTIONS:
Other: dental interproximal brush — use of this to maintain oral hygiene
  Arms: implants and oral hygiene
Other: dental floss — use of this to maintain oral hygiene
  Arms: group : implants and oral hygiene

SUMMARY:
This aim of this study is to compare different oral hygiene aids for the ability to remove plaque in patients who went through dental implant treatment and are currently on a maintenance program at the Graduate Periodontal Clinic, at the University of Manitoba, Faculty of Dentistry.

DETAILED DESCRIPTION:
Home care and Oral hygiene regimes are as well an important aspect of short and long term dental implant survival and success. The investigators profession demands us to educate the patients about the risk of peri implantitis and peri mucositis in plaque infected dentitions. In periodontal patients the areas of most ineffective plaque removal are typically the palatal/lingual and interdental areas.

there is therefore a need to developing scientific evidence to form a framework for professionals to follow when educating patients about their home care.

ELIGIBILITY:
Inclusion Criteria:

* Non smokers, with clinical probing depth around implants is less than or equal to 6mm and are currently maintained every 3 months at the graduate periodontal program

Exclusion Criteria:

* Smokers
* Probing Depth 6 or > 6mm
* Non compliant patients and patients with severe systemic conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
plaque index | one year
  plaque removal

CONTACTS AND LOCATIONS:
Overall Officials: omonkhele gertrude nwachukwu, BDS MScDPH, Principal Investigator — University of Manitoba; reem atout, DDS,DipPerio, Study Director — University of Manitoba
Locations (1):
- University of Manitoba (Graduate Periodontics Clinic), Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rasines G. The use of interdental brushes along with toothbrushing removes most plaque. Evid Based Dent. 2009;10(3):74. doi: 10.1038/sj.ebd.6400666. PMID 19820738
- [Background] Slot DE, Dorfer CE, Van der Weijden GA. The efficacy of interdental brushes on plaque and parameters of periodontal inflammation: a systematic review. Int J Dent Hyg. 2008 Nov;6(4):253-64. doi: 10.1111/j.1601-5037.2008.00330.x. PMID 19138177
- [Background] Loos B, Claffey N, Egelberg J. Clinical and microbiological effects of root debridement in periodontal furcation pockets. J Clin Periodontol. 1988 Aug;15(7):453-63. doi: 10.1111/j.1600-051x.1988.tb01600.x. PMID 3053787
- [Background] Loos B, Nylund K, Claffey N, Egelberg J. Clinical effects of root debridement in molar and non-molar teeth. A 2-year follow-up. J Clin Periodontol. 1989 Sep;16(8):498-504. doi: 10.1111/j.1600-051x.1989.tb02326.x. PMID 2778083